CLINICAL TRIAL: NCT04435132
Title: Robotic-assisted Percutaneous Access: Interventional, Non-randomized, Open-label, Non-comparative and First-in-Man Study
Brief Title: Robotic-assisted Percutaneous Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NDR Medical Technology Pte Ltd (Industry)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NDR-RA-PA-MY
Record Dates: First submitted 2020-06-09; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Kidney Stone
Keywords: PCNL; Percutaneous nephrolithotomy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Recruitment was carried out in University Malaya Medical Centre (UMMC) Hospital clinics and impatient wards. 5 patients were recruited with no preferred selection for gender or race. Patients recruited were set to be between 21 to 75 years of age.
  Patients presenting to to clinic or admitted to ward for renal stone disease were assessed for indications of PCNL. Patients were assessed for renal stone disease as per standard of care - imaging study with CT scan, renal function, clinical assessment of fitness and suitability for prone PCNL.
  Once patients were planned for prone PCNL, they will be informed about this study, the use of robotic device, potential benefits and complications by study investigators. If they are agreeable to informed consent, they will be recruited into the study.
Masking Description: Patients will undergo prone PCNL under fluoroscopic guidance and with the aid of the robotic device. They will then be admitted to inpatient ward as per standard of care for PCNL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCNL with the aid of the robotic device (Experimental): Patients will undergo prone PCNL under fluoroscopic guidance and with the aid of the robotic device.
  Interventions: Device: PCL under fluoroscopy with the aid of the robotic device

INTERVENTIONS:
Device: PCL under fluoroscopy with the aid of the robotic device — During the surgery, the robot was positioned over the estimated insertion point. It was aligned to be parallel to the fluoroscope imaging plane as much as possible. The needle is to be placed through the holder, and slightly penetrate the surface of the skin. An x-ray image is then taken to ensure that the whole device can be seen on the screen. Image calibration is then performed through the software GUI. After which, the clinician is also to perform needle tip selection. After which, needle alignment will then be performed. Once needle alignment is complete, the clinician will then advance the trocar needle into the patient's body, using the fluoroscopy to judge the penetration depth. Once the target has been reached, the needle style is to be extracted. The indication of leakage of fluid through the outer needle confirms the success of the procedure.

SUMMARY:
This is a first-in-man (FIM) study to show feasibility and safety profile of the newly developed robotic device for percutaneous access in PCNL surgery. Patients with renal stone disease who had standard indications for prone PCNL were included in the study. PCNL was conducted with percutaneous puncture with the aid of robotic device with the use of intra-operative fluoroscopy. 5 patients were recruited in this pilot study over a period of 3 months. Punctures were performed by the board-qualified urologist.

DETAILED DESCRIPTION:
All patients underwent preoperative investigations and imaging study (CT Urogram/Intravenous Pyelography) done prior to the operation as per standard operation preparation. Intraoperatively fluoroscopic imaging was done for the patients and the images were synchronized to the software. Robotic arm was placed on the site of surgery as for prone PCNL and diaphragm of the arm was centred over the site of desire calyx of entry. A needle was engaged into the centre of the diaphragm and using the software the need was aligned in the line of puncture automatically based on the fluoroscopic images. After the alignment was done the needle was advanced manually by the surgeon until the entry was confirmed by efflux of urine from the puncture needle. After the entry was confirmed a standard PCNL using 24 F or 30 F Balloon dilator was performed and stone cleared using Cyberwand/ Shockpulse etc. All the intraoperative and perioperative parameters as mentioned in the data collection form was measured. Results was analysed with the main focus on time of obtaining the puncture, accuracy of puncture, radiation exposure time till calyceal entry which was confirmed by free flow of urine and for any complications.

Patients aged between 21 to 75 years old who were diagnosed with kidney stone diseas and planned for prone PCNL with indication for surgery as per standard of care were recruited. They understood the purpose of testing and offered their voluntary and informed consent.

The robotic device i.e. ANT lesses the learning curve of percutaneous access as it reduces the need for surgeon's visualization of the calyceal system and the needle alignment. It also improved efficiency as there is less dependence on human skills during the procedure. As a whole, the FIM trial was a success. The performance of the ANT system during the trial was satisfactory. The robot alignment time is less than 30 seconds. Total puncture time was around 6 minutes and no AEs were reported.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 to 75 years
* Diagnosed with kidney stone disease and planned for prone PCNL with indication for surgery as per standard of care
* Subject who understand the purpose of testing, voluntary and informed consent, patients undergoing invasive imaging follow-up.

Exclusion Criteria:

* Bleeding disorders
* Patient on anticoagulation/antiplatelets drugs
* Pyonephrosis
* Pregnant women
* Not able to have prone position for the procedure due to comorbidities
* Moderate to severe renal failure
* The patient's life expectancy is less than 12 months
* Poor compliance and patients unable to complete the study in accordance with the requirements.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Needle insertion time | During procedure
  Time taken for PCNL procedure
Needle alignment time | During procedure
  Time taken for needle alignment
Time to target | During procedure
  Time taken for the needle to reach the calyx, from on the skin to successful needle targeting
Number of needle insertion attempts to obtain access | During procedure
  Number of attempts before successfully reaching the calyx
Radiation dosage from placement of robot to efflux of urine | During procedure
  A measure of the radiation exposed during the surgical procedure
Radiation dosage from placement of robot to successful needle target via image confirmation | During procedure
  A measure of the radiation exposed during the surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mozer P, Troccaz J, Stoianovici D. Urologic robots and future directions. Curr Opin Urol. 2009 Jan;19(1):114-9. doi: 10.1097/MOU.0b013e32831cc1ba. PMID 19057227
- [Background] Cinquin P. How today's robots work and perspectives for the future. J Visc Surg. 2011 Oct;148(5 Suppl):e12-8. doi: 10.1016/j.jviscsurg.2011.08.003. Epub 2011 Oct 5. No abstract available. PMID 21981795
- [Result] Oo MM, Gandhi HR, Chong KT, Goh JQ, Ng KW, Hein AT, Tan YK. Automated Needle Targeting with X-ray (ANT-X) - Robot-assisted device for percutaneous nephrolithotomy (PCNL) with its first successful use in human. J Endourol. 2021 Jun;35(6):e919. doi: 10.1089/end.2018.0003. PMID 29699415
- See also: Urologic robots and future directions — http://doi.org/10.1097/MOU.0b013e32831cc1ba
- See also: How today's robots work and perspectives for the future. J Visc Surg. 2011 — http://doi.org/10.1016/j.jviscsurg.2011.08.003